CLINICAL TRIAL: NCT03175159
Title: Integrated Behavioral Activation and HIV Risk Reduction Counseling for Men Who Have Sex With Men (MSM) With Stimulant Abuse
Brief Title: Integrated BA and HIV RR Counseling for MSM With Stimulant Abuse
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of California, Los Angeles (Other)
Collaborators: University of Miami (Other); The Fenway Institute (Other); Brown University (Other)
Responsible Party: Principal Investigator, Matthew Mimiaga, ScD, MPH, MA, Principal Investigator, University of California, Los Angeles
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Prevention
Other Study IDs: 1R01DA042805-01A1 (NIH)
Record Dates: First submitted 2017-06-01; First posted 2017-06-05 (Actual); Last update posted 2024-07-25 (Actual); Status verified 2024-07

CONDITIONS: Stimulant Abuse; HIV Prevention; Substance Abuse
Keywords: Risk Reduction; Crystal Methamphetamine; Cocaine; Stimulant Abuse; HIV; Behavioral Activation
MeSH Terms: conditions — Substance-Related Disorders; Risk Reduction Behavior | interventions — Standard of Care

STUDY DESIGN:
Intervention Model Description: Two-arm RTC, equally randomized between two arms: (1) the Project IMPACT intervention, "BA-RR" (behavioral activation and HIV risk reduction) counseling, which lasts ten sessions; and (2) the standard of care comparison condition, including two equivalent sexual risk reduction counseling sessions.
Who Masked: Outcomes Assessor
Masking Description: The outcome assessor will not be aware of the intervention assignment.
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Standard of Care (SOC) (Active Comparator): Sexual risk-reduction counseling sessions.
  Interventions: Behavioral: Standard of Care
- Behavioral Activation & Risk Reduction Counseling (Experimental): Behavioral activation with risk reduction counseling.
  Interventions: Behavioral: IMPACT

INTERVENTIONS:
Behavioral: IMPACT — Ten counseling sessions
  Arms: Behavioral Activation & Risk Reduction Counseling
Behavioral: Standard of Care — Two counseling sessions
  Arms: Standard of Care (SOC)

SUMMARY:
This study seeks primarily to test, in a two-arm randomized controlled trial (RCT), the efficacy of Project IMPACT, an intervention that integrates Behavioral Activation (BA) with HIV risk reduction (RR) counseling for HIV-uninfected men who have sex with men (MSM) with stimulant use disorder at risk for HIV via sexual behavior. HIV-uninfected MSM with a diagnosis of stimulant use disorder will be equally randomized to one of two study arms: (1) the Project IMPACT intervention, BA-RR counseling, which lasts ten sessions; and (2) the standard of care (SOC) comparison condition, including two equivalent sexual risk-reduction counseling sessions. Participants will be followed for one year post-randomization, with assessments at months four, eight, and 12.

DETAILED DESCRIPTION:
Project IMPACT targets both stimulant use and sexual risk reduction in effort to help individuals relearn how to enjoy safe but pleasurable activities. The intervention integrates BA, an evidence-based cognitive behavior therapy for improving mood and increasing activity, incorporated with RR counseling aimed to reduce risky sexual practices, and potential HIV acquisition. This RCT is a two-arm efficacy trial, comparing the Project IMPACT Intervention with a SOC arm. All participants will receive HIV testing, pre-/post-test risk reduction counseling, oral swab toxicology test at baseline and 12 months, assessment of interest/indication for Pre-Exposure Prophylaxis (PrEP) per Center for Disease Control guidelines, and active referral to local PrEP services as standard-of-care. Finally, the RCT will integrate resource utilization and cost-effectiveness analyses to examine cost efficiency of the Project IMPACT Intervention as a component of data analysis.

ELIGIBILITY:
Inclusion Criteria:

* Age 18 or older
* Assigned male at birth
* HIV-uninfected verified via rapid HIV test
* Self-reports in the past four months: CAS receptive or insertive with a cisgender male sexual partner, while using stimulants and without the protection of Pre-Exposure Prophylaxis (PrEP)*
* Able to read, speak, and understand English
* Willing and able to provide informed consent

Exclusion Criteria:

* Does not live in the greater Boston or Miami areas, or will move away from Boston or Miami within the next 12 months
* Self-reports being 100% adherent to PrEP in the last four months
* Unable to provide informed consent due to severe mental or physical illness, or substance intoxication at the time of interview
* Discovery of active suicidal ideation at the time of interview (participants will be referred immediately for treatment, but may join the study once resolved)-
* Involvement in any other HIV Prevention study that may interfere with the ability to test major study outcomes (e.g. another sexual risk reduction intervention or PrEP adherence intervention)

Min Age: 18 Years | Sex: Male | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Gender Based: Yes — Intervention addresses stimulant use and HIV risk reduction in MSM
Enrollment: 205 (Actual)
Dates: Start 2018-03-01 (Actual); Primary Completion 2024-03-01 (Actual); Study Completion 2024-03-01 (Actual)

PRIMARY OUTCOMES:
Reduction in Condomless Anal Sex Acts (CAS) over study follow-up | Baseline, 4 month, 8 month, 12 month
  A self reported change in the number of CAS with men without protection of PrEP

SECONDARY OUTCOMES:
Reduction in the number of stimulant use episodes over study follow-up | Baseline, 4 month, 8 month, 12 month
  A self reported change in the number of stimulant use episodes over study follow-up

CONTACTS AND LOCATIONS:
Overall Officials: Matthew J Mimiaga, ScD, MPH, Principal Investigator — University of California, Los Angeles, Fielding School of Public Health; Steve Safren, PhD, Principal Investigator — University of Miami
Locations (2):
- United States (2):
  - University of Miami, Miami, Florida
  - Fenway Community Health Center, Boston, Massachusetts

IPD SHARING:
Plan to Share IPD: Yes
Raw data for additional analysis will be available to outside individuals through contacting the Multiple Principal Investigators (MPI) at two different times. The first will be after all of the baseline data is collected. We will institute a concept plan process where internal study staff first have the availability to write papers or give presentations on particular topics. After this, if outside individuals wish to analyze data, we will welcome this collaboration. A similar process will happen for outcome data; however, this will not be possible until the publication and release of the outcome paper(s). The MPIs (Mimiaga and Safren) will store the data indefinitely and allow access for pooled data analysis projects, or projects for outside individuals. Information regarding the availability of data for analysis will be listed on the MPIs' program's web page. Contact information for the MPIs will be listed in all manuscripts and publications as another means to access data.
Time Frame: The first time point at which outside investigators may request IPD will be after all of the baseline data has been collected and internal study staff have been offered the availability to write papers or give presentations on particular topics. A similar process will take place for outcome data following publication and release of the outcome paper(s). The MPIs (Mimiaga and Safren) will store the data indefinitely.
Access Criteria: Raw data for additional analysis will be available to outside individuals through contacting the Multiple Principal Investigators (MPI). We will institute a concept plan process where internal study staff first have the availability to write papers or give presentations on particular topics. After this, if outside individuals wish to analyze data, we will welcome this collaboration. The MPIs (Mimiaga and Safren) will store the data indefinitely and allow access for pooled data analysis projects, or projects for outside individuals. Information regarding the availability of data for analysis will be listed on the MPIs' program's web page.

REFERENCES:
- [Derived] Klasko-Foster LB, Biello KB, Lodge W 2nd, Olson J, Mimiaga MJ. Transitioning from Face to Face to the Digital Space: Best Practices and Lessons Learned Leveraging Technology to Conduct HIV-Focused Interventions. Telemed J E Health. 2022 Jul;28(7):1070-1073. doi: 10.1089/tmj.2021.0190. Epub 2022 Jan 6. PMID 34995162
- [Derived] Mimiaga MJ, Pantalone DW, Biello KB, Glynn TR, Santostefano CM, Olson J, Pardee DJ, Hughto JMW, Garcia Valles J, Carrico AW, Mayer KH, Safren SA. A randomized controlled efficacy trial of behavioral activation for concurrent stimulant use and sexual risk for HIV acquisition among MSM: project IMPACT study protocol. BMC Public Health. 2018 Jul 25;18(1):914. doi: 10.1186/s12889-018-5856-0. PMID 30045702

DOCUMENTS (1):
  • Informed Consent Form (2021-11-09): https://cdn.clinicaltrials.gov/large-docs/59/NCT03175159/ICF_002.pdf